CLINICAL TRIAL: NCT00109304
Title: Safety, Tolerability and Immunogenicity of the Venezuelan Equine Encephalitis (VEE) Attenuated Live-Virus Vaccine VEE IA/B V3526 in VEE-Naive Healthy Volunteers After Single Dose Subcutaneous Administration
Brief Title: Safety, Tolerability and Immunogenicity of the Venezuelan Equine Encephalitis (VEE) Attenuated Live-Virus Vaccine
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: DynPort Vaccine Company LLC, A GDIT Company (Industry)
Responsible Party: Dr. K. McKee, Chief Medical Officer, DynPort Vaccine Company
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: VEE-01
Record Dates: First submitted 2005-04-27; First posted 2005-04-27 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Venezuelan Equine Encephalitis
Keywords: Venezuelan Equine Encephalitis; VEE; Vaccine; Provide protective immunity against VEE subtypes IA/B
MeSH Terms: conditions — Encephalomyelitis, Venezuelan Equine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: VEE 3526

SUMMARY:
This study is being done to determine the safety and tolerability of a new investigational vaccine referred to as VEE IA/B V3526, which may induce production of specific antibodies in vaccinated humans, and may protect them against infection with the Venezuelan Equine Encephalitis (VEE) Virus.

DETAILED DESCRIPTION:
Safety Objectives: 1) To determine preliminary safety, reactogenicity, and tolerability of VEE IA/B V3526 in VEE-naïve healthy volunteers after single dose subcutaneous (SC) administration; 2) To evaluate virological safety by assessing serum viremia and viral shedding in nose and throat.

Immunogenicity Objectives: 1) To assess the humoral immune response (plaque reduction neutralizing antibody titer (PRNT)) against VEE subtype IA/B after SC administration of different dose-levels of the VEE IA/B V3526 vaccine candidate; 2) To assess duration of immune response over six months after the VEE IA/B V3526 vaccination based on PRNT; and 3) To identify two suitable VEE IA/B V3526 vaccine dose-levels for future administration in dose optimization and expanded safety studies.

Exploratory Objectives: 1) To collect and store serum for future development of immunogenicity assays (e.g., ELISA) against multiple VEE subtypes IA/B, IE, IIIA, and other possible subtypes; 2) To collect and store serum for future use in the development of a passive transfer challenge model; 3) Collect VEE IA/B V3526 positive serum (Positive Control Serum) at the Day 21 visit.

ELIGIBILITY:
Inclusion Criteria:

* The volunteer is a male or female between 18 and 40 years of age (inclusive).
* The volunteer is able and willing to comply with the protocol procedures: 2-week 15 nights/ (14-day) in-patient stay and availability for follow-up visits for six months post vaccination.
* The volunteer is in good health, as determined by the Investigator following a complete medical history and physical examination, and the volunteer has had no clinically significant illness by medical history or exam (e.g., asthma, hypertension) or requiring hospitalization within the six months before vaccination in this study.
* The volunteer has the following laboratory parameters within normal range: *total WBC, *hemoglobin, *platelets, *LFT (liver function tests (AST, ALT, ALP, bilirubin) and *negative for proteinuria. Other laboratory parameters must be within 10% of the upper or lower limits of the normal range of the Northwest Kinetics clinical laboratory and not clinically significant as assessed by the Investigator and/or Sponsor Medical Monitor.
* Female volunteers must not be pregnant or nursing, or must be of non-childbearing potential (e.g., surgically sterilized or postmenopausal). If volunteers are women of childbearing potential (WCBP), they must verbalize use of an acceptable method of contraception (i.e., hormonal contraception (injectable or oral) or intrauterine device) or abstinence for at least 30 days before and through 180 days after vaccination.
* The volunteer agrees not to donate blood for at least six months after vaccination.
* The volunteer has successfully completed the Test of Understanding for the protocol (answered 90% questions correctly), has signed an ICF (inclusive of the HIPAA authorization).
* The volunteer agrees to have his/her blood samples collected and stored for future investigations related to VEE vaccine development (e.g., assay development) and future VEE-related research studies.
* The volunteer has been provided Northwest Kinetics Site Subject Instructions for participation and agrees with the Northwest Kinetics Site Subject Instructions.

Exclusion Criteria:

* History of exposure to VEE, WEE (Western Equine Encephalitis), EEE (Eastern Equine Encephalitis), and/or CHIK (Chikungunya) with or without serological evidence (PRN).
* History of allergic reaction to human serum albumin (HSA) or other vaccine components (i.e., DMEM), or history of anaphylaxis or serious adverse reactions to other vaccines.
* History of seizure disorder or history of encephalitic process with sequelae.
* Frequent or severe headaches of any etiology.
* Chronic, severe, or recurrent joint pain or arthritis of any etiology.
* History of diabetes in first degree relatives.
* History of gestational diabetes.
* Abnormal fasting blood glucose.
* Current use of antiviral and other systemic immunomodulatory pharmacotherapy. Use of immunosuppressive agents or corticosteroids (i.e., systemic total dose of 20 mg/day or 2 mg/kg or 20 mg/day, "burst" therapy, intra-nasally administered, or inhaled steroids within the 3 months prior to the study).
* Currently enrolled in an investigational protocol or has participated in any clinical trial using an investigational product within the last month.
* Current or planned participation in a blood donation resulting in a blood volume of > 450 mL per 8 week period.
* Vaccination with any attenuated live-vaccine (e.g., varicella-zoster vaccine) within 60 days prior to test-vaccine administration.
* Vaccination with any inactivated vaccine (e.g., polio or hepatitis A vaccine) within 30 days prior to test-vaccine administration.
* Oral temperature >100.0°F at the time of scheduled test-vaccine administration.
* The volunteer has a clinically significant abnormality on the ECG.
* The volunteer has a body mass index >= 40 kg/m2 or is greater than or equal to 100 lbs over the ideal body weight.
* Personal or family history of multiple sclerosis, as immune system stimulation may exacerbate this disorder.
* Signs or symptoms of illness at the time of scheduled test-vaccine administration, which are considered clinically relevant by the Principal Investigator (PI, Study Doctor).
* WCBP with current or planned pregnancy within 30 days before scheduled test-vaccine administration and/or during the study (i.e., Day 0 through Day 180). Female volunteer (WCBP) is pregnant, breastfeeding, tests positive on a pregnancy test any time before vaccination, or is unwilling to use an acceptable method of contraception (i.e., hormonal contraception (injectable or oral) or intrauterine device) or abstinence within 30 days before and during the 180 days of the study.
* Positive HIV, HBsAg or HCV serology.
* The volunteer has a positive result on a urine drug screen that tests for common substances of abuse such as amphetamines, barbiturates, benzodiazepines, cocaine, opiates, and cannabinoids. (If positive on screen, confirmatory testing shall be performed where applicable).
* The volunteer has a previous diagnosis of any serious psychiatric disorder. For this purpose, serious psychiatric disorder is defined as illness requiring hospitalization within previous 12 months and/or routine administration of more than one medication to control anxiety, mood, or sleep disorder; or history of suicide attempt.
* The volunteer is considered, for any reason, by the Investigator to be an unsuitable candidate for receipt of an investigational treatment. The specific reason for exclusion under this element must be completely documented in the screening case report form.
* The volunteer is unwilling to comply with all aspects of the protocol through the post vaccination Day 180 (±7 days) assessment, or the volunteer's medical or psychiatric condition or occupational responsibilities preclude compliance with the protocol-specified procedures.
* The volunteer has screening laboratory values for total WBC, Hemoglobin, platelets, LFT (AST, ALT, ALP, Bilirubin) that are not within normal range and/or a positive urine test for proteinuria.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2005-07; Study Completion 2006-12

PRIMARY OUTCOMES:
Incidence and character of adverse events considered related to the VEE IA/B V3526 vaccine
Level and duration of serum viremia and viral shedding in nose and/or throat

SECONDARY OUTCOMES:
Store samples collected for future use in the development of immunogenicity assays against multiple VEE subtypes IA/B, IE, IIIA, and other possible subtypes
Store samples collected for the future development of the passive transfer challenge model
Store VEE IA/B V3526 Positive Control Serum to be used in future studies

CONTACTS AND LOCATIONS:
Locations (1):
- Northwest Kinetics, Inc., Tacoma, Washington, United States